CLINICAL TRIAL: NCT02052674
Title: Retained Urine Volume and Bacteriuria in Traditional Versus Vented Urine Drainage Systems
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to enroll any patients in the study due to other on-going studies.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201300634
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Bacteriuria
Keywords: Precursor to CAUTI
MeSH Terms: conditions — Bacteriuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vented urinary drainage system (Experimental): This group will be catheterized with a vented urinary drainage system. Several data sets will be evaluated to compare the two arms of the study: retained urine volume, the difference (ΔH) in meniscus heights in the dependent loops, time necessary for drainage of dependent loops, and incidence of bacteriuria.
  Interventions: Device: Vented urinary drainage system
- Non-vented urinary drainage system (Active Comparator): This group will be catheterized with a non-vented urinary drainage system. Several data sets will be evaluated to compare the two arms of the study: retained urine volume, the difference (ΔH) in meniscus heights in the dependent loops, time necessary for drainage of dependent loops, and incidence of bacteriuria.
  Interventions: Device: Non-vented urinary drainage system

INTERVENTIONS:
Device: Vented urinary drainage system — This group will be catheterized with a vented urinary drainage system. Several data sets will be evaluated to compare the two arms of the study: retained urine volume, the difference (ΔH) in meniscus heights in the dependent loops, time necessary for drainage of dependent loops, and incidence of bacteriuria.
  Other Names: Covidien vented foley catheter; TopVent; Covidien Dover Precision Premium Drainage bag
  Arms: Vented urinary drainage system
Device: Non-vented urinary drainage system — This group will be catheterized with a non-vented urinary drainage system. Several data sets will be evaluated to compare the two arms of the study: retained urine volume, the difference (ΔH) in meniscus heights in the dependent loops, time necessary for drainage of dependent loops, and incidence of bacteriuria.
  Other Names: Bard urine drainage system; Conventional catheter; Bard Silver-Coated
  Arms: Non-vented urinary drainage system

SUMMARY:
The purpose of this study is to see if there are differences in urine drainage between two types of indwelling bladder catheter systems (Foley catheter) in hospitalized patients. The difference between the two catheters is that one catheter is vented (the study catheter) and the other is a standard non-vented catheter. The vented catheter may drain urine better than a standard non-vented catheter.

If a vented catheter drains the bladder better than a non-vented catheter it may lower the risk of retained urine in the bladder which could help prevent urinary tract infections.

DETAILED DESCRIPTION:
During hospitalization, while in the surgical intensive care unit beginning the day after surgery, measurements of the subject's urine drainage system will be taken at daily study visits: retained urine volume, dependent loops, incidence of bacteriuria, and thigh diameter.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a planned surgery
* Anticipated indwelling bladder catheter placement for greater than 24 hours
* Anticipated post-op admission to a surgical ICU

Exclusion Criteria:

* Unstable renal function as self-reported
* Anticipated bandaged postoperative suprapubic incisions
* Anatomical deformity that precludes appropriate suprapubic access for ultrasound bladder scanning
* Surgical procedure that prevents accurate core body temperature by any means other than by bladder temperature

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Bacteriuria | 7 days
  Evidence of bacteriuria, a potential precursor to Catheter Associated Urinary Tract Infection (CAUTI), will be used to study the potential effect of the vented urinary drainage system intervention on CAUTI.

SECONDARY OUTCOMES:
Retained Urine | 7 days
  One potential source for the risk of developing a Urinary Tract Infection (UTI) is related to residual urine volume in the bladder
Presence of biofilms in catheter materials | 7 days
  A key contributor to bacteriuria is formation of biofilms in the catheter and catheter tubing.

CONTACTS AND LOCATIONS:
Overall Officials: William B. Smith, MD, Principal Investigator — University of Florida